CLINICAL TRIAL: NCT05053711
Title: Augmented Efficacy of Repetitive Peripheral Magnetic Stimulation on the Repetitive Transcranial Magnetic Stimulation on Upper Limb Function in Patients With Stroke: a Randomized Controlled Trial
Brief Title: Augmented Efficacy of rPMS on the rTMS on Upper Limb Function in Patients With Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 202002582A3
Record Dates: First submitted 2021-09-03; First posted 2021-09-22 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2021-08

CONDITIONS: Stroke
Keywords: Repetitive transcranial magnetic stimulation; Repetitive peripheral magnetic stimulation; stroke; novel treatment
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- rTMS+rPMS_iTBS_M (Experimental): In this group, they received iTBS on affected hemisphere after following iTBS at median nerve on affected hand.
  Interventions: Device: rTMS+rPMS_iTBS_M
- rTMS+rPMS_cTBS_M (Experimental): In this group, they received iTBS on affected hemisphere after following cTBS at median nerve on affected hand.
  Interventions: Device: rTMS+rPMS_cTBS_M
- rTMS+sham rPMS_M (Sham Comparator): In this group, they received iTBS on affected hemisphere after following sham TBS stimulation at median nerve on affected hand.
  Interventions: Device: rTMS+sham rPMS_M
- rTMS+rPMS_iTBS_U (Experimental): In this group, they received iTBS on affected hemisphere after following iTBS at ulnar nerve on affected hand.
  Interventions: Device: rTMS+rPMS_iTBS_U
- rTMS+rPMS_cTBS_U (Experimental): In this group, they received iTBS on affected hemisphere after following cTBS at ulnar nerve on affected hand.
  Interventions: Device: rTMS+rPMS_cTBS_U
- rTMS+sham rPMS_U (Sham Comparator): In this group, they received iTBS on affected hemisphere after following sham TBS stimulation at ulnar nerve on affected hand.
  Interventions: Device: rTMS+sham rPMS_U

INTERVENTIONS:
Device: rTMS+rPMS_iTBS_M — Repetitive peripheral magnetic stimulation (rPMS) intermittent theta-burst stimulation pattern (iTBS) will intermittently give a 2 s train of iTBS every 10s repeated 2 times for a total of 40 times at median nerve on the affected hand(low pulse: 1200 pulses in total). Then following Repetitive transcranial magnetic stimulation (rTMS) will intermittently give a 2 s train of iTBS every 10s repeated 2 times for a total of 40 times on affected hemisphere(low pulse: 1200 pulses in total).
  Arms: rTMS+rPMS_iTBS_M
Device: rTMS+rPMS_cTBS_M — Repetitive peripheral magnetic stimulation (rPMS) continuous burst stimulation pattern (cTBS) will intermittently give a cTBS treatment consists of a continuous train of TBS for 40 seconds repeated for 2 times at median nerve on the affected hand(low pulse: 1200 pulses in total). Then following Repetitive transcranial magnetic stimulation (rTMS) will intermittently give a 2 s train of iTBS every 10s repeated 2 times for a total of 40 times on affected hemisphere(low pulse: 1200 pulses in total).
  Arms: rTMS+rPMS_cTBS_M
Device: rTMS+sham rPMS_M — Repetitive peripheral magnetic stimulation (rPMS) sham burst stimulation pattern (sham TBS) will intermittently give a sham TBS treatment consists of a continuous train of TBS for 40 seconds at median nerve on the affected hand(almost no pulse: 1200 pulses in total). Then following Repetitive transcranial magnetic stimulation (rTMS) will intermittently give a sham TBS treatment consists of a continuous train of TBS for 40 seconds on affected hemisphere(almost no pulse: 1200 pulses in total).
  Arms: rTMS+sham rPMS_M
Device: rTMS+rPMS_iTBS_U — Repetitive peripheral magnetic stimulation (rPMS) intermittent theta-burst stimulation pattern (iTBS) will intermittently give a 2 s train of iTBS every 10s repeated 2 times for a total of 40 times at ulnaris nerve on the affected hand(low pulse: 1200 pulses in total). Then following Repetitive transcranial magnetic stimulation (rTMS) will intermittently give a 2 s train of iTBS every 10s repeated 2 times for a total of 40 times on affected hemisphere(low pulse: 1200 pulses in total).
  Arms: rTMS+rPMS_iTBS_U
Device: rTMS+rPMS_cTBS_U — Repetitive peripheral magnetic stimulation (rPMS) continuous burst stimulation pattern (cTBS) will intermittently give a cTBS treatment consists of a continuous train of TBS for 40 seconds repeated for 2 times at ulnar nerve on the affected hand(low pulse: 1200 pulses in total). Then following Repetitive transcranial magnetic stimulation (rTMS) will intermittently give a 2 s train of iTBS every 10s repeated 2 times for a total of 40 times on affected hemisphere(low pulse: 1200 pulses in total).
  Arms: rTMS+rPMS_cTBS_U
Device: rTMS+sham rPMS_U — Repetitive peripheral magnetic stimulation (rPMS) sham burst stimulation pattern (sham TBS) will intermittently give a sham TBS treatment consists of a continuous train of TBS for 40 seconds at ulnar nerve on the affected hand(almost no pulse: 1200 pulses in total). Then following Repetitive transcranial magnetic stimulation (rTMS) will intermittently give a sham TBS treatment consists of a continuous train of TBS for 40 seconds on affected hemisphere(almost no pulse: 1200 pulses in total).
  Arms: rTMS+sham rPMS_U

SUMMARY:
Repetitive transcranial magnetic stimulation (rTMS) and repetitive peripheral magnetic stimulation (rPMS) are innovative treatments for patients with stroke. Therefore, augmented efficacy of rPMS on the rTMS is employed in this project. This proposal aims at exploring different novel treatment strategies in the treatment of UE dysfunction in patients with stroke: augmented efficacy of rPMS on the rTMS. Several aims in this study include (1) identifying the most optimal treatment protocols for rPMS (TBS treatment and nerve stimulation location), (2 ) establish a novel treatment protocol (augmented efficacy of rPMS on the rTMS), (3) identifying augmented efficacy of rPMS on the rTMS, (4) determining the mechanism of neuro-motor control, and (5) related biomarkers for the novel treatment protocol. The investigators applied a 3-year plan before, however, the Ministry of Science and Technology plan passed one year only (108-2314-B-182-043-). The investigators carried out the pilot study to investigate the augmented effects of rPMS (radial nerve) on the rTMS in the treatment of upper limb function in patients with stroke patients. The previous plan had preliminary results. This year the investigators will apply for a three-year plan to continue the previous pilot study for getting the comprehensive results.

DETAILED DESCRIPTION:
This study intends to further explore whether rPMS intervention in different nerves can augment rTMS efficacy on upper limb function in patients with stroke. A total of 72-96 patients with stroke will be recruited in 2 phases and 36-48 participants will be divided into four groups according to their severity and the onset of stroke, and then randomly enrolled into 3 groups in each phase (12-16 participants in each group) based on different rPMS- stimulated methods and location. All patients will receive the rPMS in addition rTMS on the brain cortex. In phase 1, each patient will receive either one of three rPMS methods on median nerve (iTBS, cTBS, sham). During phase 2, each patient will receive either one of three rPMS methods on ulnar nerve. Outcome measures include clinical assessments based on International Classification of Functioning, Disability and Health (ICF) and motor control (Motor Evoked Potential, MEP, kinetics, and kinematics) that administered at pretest, posttest, and 3-month follow-up. This study aims to establish a novel assessment and treatment protocols in patients with stroke. The intervention will be conducted 10 times for each participant. The optimal effective treatment protocol of augmented efficacy of rPMS on the rTMS will also be established. The results of this study will be applied to the translational and evidence-based medicine of the neuro-rehabilitation field of stroke research.

ELIGIBILITY:
Inclusion Criteria:

* first stoke and in stable phase
* age 20-80 years
* unilateral brain lesions with unilateral hemiplegia
* brain wave examination without epileptic waves

Exclusion Criteria:

* brain stem or cerebellar stroke
* Patients with epilepsy
* Patients with aneurysm or cerebrovascular malformation
* Patients with mental illness
* Patients with degenerative diseases (such as neurodegenerative diseases)
* Patients with severe intelligence or language barriers (such as mental retardation or severe communication impairment)
* Patients with serious medical conditions (such as heart failure)
* Patients with acute disease (such as infection)
* Patients had metal implants in the body (such as cardiac rhythm or brain metal implants, metal clips for aneurysms)
* Patients had botox injection or surgery in the first half of the study
* Pregnant woman or breastfeeding woman
* other obstacles (such as claustrophobia, obesity, etc.)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Motion analysis at after treatment and three month | baseline, after two weeks of treatment, 3 months
  All participants will be instructed to perform a series of upper-extremity tasks. The tasks include reaching and grasping. An 7-camera motion analysis system (Vicon system, 3-D Oxfort Metrics Ltd, Oxford, UK) is used in conjunction with a personal computer to capture the movement of markers placed on the participant's body; analog signals were collected simultaneously. Movements were recorded at 120 Hz and digitally low-pass filtered at 5 Hz using a second-order Butterworth filter. Reference markers are placed on the distal interphalangeal joints of the thumb and index finger, the styloid process of the ulna, proximal end of the second metacarpal, and the object.
Change from baseline Motor evoked potential at afte treatment and three month | baseline, after two weeks of treatment, 3 months
  The comparison of baseline of Motor Evoked Potential for stroke after different therapy, including resting motor threshold (RMT), active motor thresholds (AMT), input-output curve (IO curve) and stationary period.
Change from baseline Myoton at after treatment and three month | baseline, after two weeks of treatment, 3 months
  The comparison of baseline of Myoton for stroke after different therapy, assessing the functional status of skeletal muscle, including tone or state of tension(natural oscillation frequency[Hz]), biochanical properties(dynamic stiffness [N/m], logarithmic decrement of natural oscillation), viscoelastic properties(mechanical stress relaxation time [ms], ratio of deformation and relaxation time, characterising Creep (Deborah number)).
Change from baseline Muscle strength at after treatment and three month | baseline, after two weeks of treatment, 3 months
  The comparison of baseline of Muscle strength for stroke after different therapy, including lateral pinch, palmar pinch, and tip pinch, the strength will be tested by hand dynamometer.
Change from baseline Brunnstrom stage at after treatment and three month | baseline, after two weeks of treatment, 3 months
  The Brunnstrom stage is used to classify the severity of stroke patient according to specific movement.
Change from baseline Fugl Meyer Assessment at after treatment and three month | baseline, after two weeks of treatment, 3 months
  The Fugl Meyer Assessment is used to measure upper and lower extremity motor , range of motion, sensation, pain and balance.
Change from baseline Modified Ashworth Scale at after treatment and three month | baseline, after two weeks of treatment, 3 months
  The Modified Ashworth Scale is used to measure the muscle tone of affected limb, for each item minimum value is 0 and maximum value is 4, higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Change from baseline Action Research Arm Test at after treatment and three month | baseline, after two weeks of treatment, 3 months
  The Action Research Arm Test is used to measure bilateral gross manual and finger dexterity.
Change from baseline Box and Block Test at after treatment and three month | baseline, after two weeks of treatment, 3 months
  The Box and Block Test (BBT) measures unilateral gross manual dexterity.
Change from baseline Nine-Hole test at after treatment and three month | baseline, after two weeks of treatment, 3 months
  The Nine-Hole Peg Test (NHPT) is used to measure finger dexterity in patients with various neurological diagnoses.
Change from baseline Jebson Taylor Hand Function Test at after treatment and three month | baseline, after two weeks of treatment, 3 months
  The Jebson Taylor Hand Function Test (JTHFT) is used to assess a broad range of unilateral hand functions required for activities of daily living(ADLs).
Change from baseline Functional Independence Measure at after treatment and three month | baseline, after two weeks of treatment, 3 months
  The purpose of Functional Independence Measure(FIM) is to understand and track adult's life function performance, progress and goal achievement. There are three main areas: self-care, mobility, and cognition. The score is from 1 to 7 points, 1 is completely dependent, and 7 is completely independent.
Change from baseline Motor Activity Log at after treatment and three month | baseline, after two weeks of treatment, 3 months
  The Motor Activity Log(MAL) is used to measure the quality and quantity of a stroke patient when performing activities using the affected hand.
Change from baseline Wolf Motor Function Test at after treatment and three month | baseline, after two weeks of treatment, 3 months
  The Wolf Motor Function Test(WMFT) is used to measure unilateral motor quality and strength.
Change from baseline Nottingham Health Profile at after treatment and three month | baseline, after two weeks of treatment, 3 months
  The Nottingham Health Profile(NHP) is a questionnaire that assesses the quality of life associated with health. There are a total of 38 items, divided into six sub-items: mobility, social isolation, emotional response, pain, sleep and energy.
Change from baseline Stroke Impact Scale at after treatment and three month | baseline, after two weeks of treatment, 3 months
  The Stroke Impact Scale(SIS) is used to measure the influence of several aspects after stroke, for each item minimum value is 1 and maximum value is 5, higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Ling Chen, Study Director — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memoria Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No